CLINICAL TRIAL: NCT02900079
Title: New Tools for Diagnosis and Management of Febrile Illness in Travelers to the Tropics: a Cohort Study- JOKA I
Brief Title: Use of Malaria Rapid Diagnostic Tests as a Decision Aid for the Management of Fever by International Travelers
Acronym: JOKA-I
Status: Withdrawn | Type: Observational
Why Stopped: delays in obtaining study materials
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Other Study IDs: B300201627244
Record Dates: First submitted 2016-03-16; First posted 2016-09-14 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Fever; Malaria
Keywords: malaria; rapid diagnostic test; travel; fever; self care
MeSH Terms: conditions — Fever; Malaria | interventions — Rapid Diagnostic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — sera, capillary blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- travelers: persons intending to travel for 3 weeks or longer to South-East Asia, Sub-Saharan Africa or South-/ Central America; they will be trained to use a rapid diagnostic test for malaria antigen when febrile. Upon a positive test result they are recommended to use standby emergency treatment (SBET)
  Interventions: Device: rapid diagnostic test for malaria antigen

INTERVENTIONS:
Device: rapid diagnostic test for malaria antigen — rapid diagnostic test for malaria antigen to be used by travelers when febrile

SUMMARY:
This study is part of a larger prospective cohort study (JOKA), designed to study the incidence and etiological spectrum of febrile illness occurring during a travel to the tropics, as well as clinical course, care, treatment and outcome of these febrile illness episodes. Its objective is to evaluate the clinical use of malaria rapid diagnostic tests (RDT) by travelers or their peers during travel, as a decision aid for the management of febrile illness in the tropics.

If the study demonstrates that malaria can be ruled out safely by travelers themselves using a RDT, a combination of self/peer testing with SBET may become an alternative to antimalarial chemoprophylaxis in travel medicine.

DETAILED DESCRIPTION:
Objectives:

To evaluate the clinical use of malaria rapid diagnostic tests (RDT) by travelers or their peers during travel, as a decision aid for the management of febrile illness.

Design: Prospective cohort study of febrile illness in international travelers

Population: Travelers who are going to destinations in the tropics (South-East Asia (SEA), Sub-Saharan Africa (SSA) and South America (SCA)) for 3 weeks or longer will be invited to participate and, after obtaining informed consent, recruited in the study protocol(s) at the time of planning departure (directly at the ITM or through travel/ humanitarian relief organizations).

Methods: Participants will be offered pre-, per- and post-travel consultation as explained below:

Inclusion through ITM; 1. Pre-travel consultation at a certified travel clinic ("Erkend Centrum voor Medisch Reisadvies en Inentingen") will systematically be recommended; this consultation will include:

(1) routine travel advice directed at travel destination, (including vaccinations and prescription for anti-malarial chemoprophylaxis according to current recommendations, details of which are published at www.reisgeneeskunde.be and (2) the following research-related activities:

* Briefing sessions on the topic "Fever in The Tropics" by an ITM physician (during this session the differences between fever at home and in the tropics will be addressed and the importance of consulting a local doctor will be stressed).
* Collection and recording of demographic, clinical and travel data.
* Sampling of a baseline serum sample (for paired pre- and post-travel diagnostic analysis).
* Training of travelers, peers and travel guides to perform and interpret a malaria RDT (training is a prerequisite for study participation).
* Provision of study materials (study diary/apps, malaria kits, thermometer, …) and written instructions for use during travel if fever occurs.

  2. During travel
* In case of any illness (associated with fever or not), the traveler will record symptoms in the study diary.
* If fever is documented (axillary temperature ≥ 37.8°C - or in case a thermometer is not immediately available, fever sensation in association with sweats or chills)- blood from a finger prick will be collected for use of the malaria rapid diagnostic test (RDT, presenting as a nitrocellulose strip in a plastic cassette).
* In case of a positive RDT result the traveler is advised to start artemisinin based combination therapy (ACT) as 'standby emergency treatment' (SBET) for malaria as soon as possible.
* All febrile travelers are advised to seek medical attendance as they would do when not participating in the study.
* To guide interpretation of the RDT test results, precise instructions will be provided (Annex); to allow post-hoc verification, photographs of the RDT test will be taken at the time of reading, to be kept or sent to the ITM study team for advice (see below)quality control and study documentation. Participants will also asked to store the RDT cassette for further analysis upon return.
* The final decision to use standby emergency treatment malaria treatment (SBET) is made by the study participant, in accordance with precise and written instructions.
* The study team (Tropical medicine experts at ITM) will be available for teleconsultation by Email or Telephone, and will provide medical advice (including assistance in RDT reading and interpretation) within 12 hours. Note: contacting the ITM study team is an option, but should not cause delay in treating suspected malaria.
* Study participants will collect all relevant data related to the (outcome of the) illness episode (duration of symptoms, consultation of a health practitioner, admission/duration of stay in a hospital, treatment received and timing, repatriation)

  3. Post-travel consultation will be scheduled for all study participants who experience(d) any illness (febrile or not) within a week after travel- sooner if the medical condition requires so- and for those who have no complaints but do seek post-travel health evaluation.
* A structured clinical evaluation will be performed by an expert in travel medicine and will be recorded in the database. Laboratory evaluation will include hematological, biochemical and microbiological/parasitological analysis
* Used RDTs will be collected for confirmation of the test result by Polymerase Chain Reaction (PCR).

  * Data analysis : All data (demographic, geographic, clinical, laboratory and final diagnosis) will be recorded in an encoded database. Descriptive and inferential statistics as appropriate, STATA 14.
  * Sample size: n= 350 fever cases; at an incidence of fever of 8% a cohort of 4400 (healthy) travelers will be recruited over 30 months (Feb 2016 - Aug 2018).
  * Endpoints:
* To determine the post-test probability for malaria after a negative RDT result (i.e. excluding power of the RDT) as well as other measures of diagnostic accuracy (sensitivity, specificity, positive predictive value) in travelers with febrile illness, when performed by travelers (or their peers)- compared with PCR detection of Plasmodium spp. on the RDT after return
* Qualitative description of ease of self-/peer- use of malaria RDT
* Incidence rates for malaria (by use of RDT and post-travel PCR on RDT)
* Clinical course and outcomes of (self-)management of febrile illness during travel.

Expected results and relevance:

If the study demonstrates that malaria can be ruled out safely by travelers themselves using a RDT, a combination of self/peer testing with SBET may become an alternative to antimalarial chemoprophylaxis in travel medicine.

ELIGIBILITY:
Inclusion Criteria:

* residing in Belgium
* Attend a briefing session on the topic "Fever in The Tropics" by an ITM physician
* able to comply with study procedures:
* carry and complete a study diary in case of illness
* be trained to use RDT
* Willing and able to provide written informed consent
* Adults fulfilling all criteria and volunteer to have their RDT collected by their trained peers during travel, may be included for analysis after obtaining informed consent upon post-travel evaluation.

Exclusion Criteria:

* known intolerance or hypersensitivity to artemisinine based combination therapy
* known pregnancy at time of travel

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: persons intending to travel to Asia, Africa, or America for a minimum duration of 3 weeks
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
negative predictive value of a malaria RDT when used by travelers with febrile illness | up to 12 weeks followup
  malaria RDT results will be compared to post hoc PCR diagnosis of malaria on the original test strip; the negative predictive value (NPV) will be calculated in a travelers' cohort. A NPV > 99,0 % will be considered as safe to rule out malaria.

SECONDARY OUTCOMES:
Qualitative description of ease of self-/peer- use of malaria RDT, measured by a self-reported questionnaire | up to 12 weeks
Time to treatment measured from time of obtaining test results by self-reporting | up to 12 weeks
  Use of study diary
Duration of symptoms by self-reporting | up to 12 weeks
  Use of study diary
Description of clinical symptoms and their frequencies by self-reporting | up to 12 weeks
  Use of study diary
self-reported management of illness in structured study diary | up to 12 weeks
  self-treatment, consultation, hospitalization
final clinical outcome of illness | up to 12 weeks
  change of travel plans, repatriation, hospitalization, death as a result of illness during travel

CONTACTS AND LOCATIONS:
Overall Officials: Jan Jacobs, MD PhD, Study Chair — Institute of Tropical Medicine, Antwerp, Belgium
Locations (1):
- ITM, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jelinek T, Schulte C, Behrens R, Grobusch MP, Coulaud JP, Bisoffi Z, Matteelli A, Clerinx J, Corachan M, Puente S, Gjorup I, Harms G, Kollaritsch H, Kotlowski A, Bjorkmann A, Delmont JP, Knobloch J, Nielsen LN, Cuadros J, Hatz C, Beran J, Schmid ML, Schulze M, Lopez-Velez R, Fleischer K, Kapaun A, McWhinney P, Kern P, Atougia J, Fry G, da Cunha S, Boecken G. Imported Falciparum malaria in Europe: sentinel surveillance data from the European network on surveillance of imported infectious diseases. Clin Infect Dis. 2002 Mar 1;34(5):572-6. doi: 10.1086/338235. Epub 2002 Jan 21. PMID 11803507
- [Background] Checkley AM, Smith A, Smith V, Blaze M, Bradley D, Chiodini PL, Whitty CJ. Risk factors for mortality from imported falciparum malaria in the United Kingdom over 20 years: an observational study. BMJ. 2012 Mar 27;344:e2116. doi: 10.1136/bmj.e2116. PMID 22454091
- [Background] Seringe E, Thellier M, Fontanet A, Legros F, Bouchaud O, Ancelle T, Kendjo E, Houze S, Le Bras J, Danis M, Durand R; French National Reference Center for Imported Malaria Study Group. Severe imported Plasmodium falciparum malaria, France, 1996-2003. Emerg Infect Dis. 2011 May;17(5):807-13. doi: 10.3201/eid1705.101527. PMID 21529388
- [Background] Landry P, Iorillo D, Darioli R, Burnier M, Genton B. Do travelers really take their mefloquine malaria chemoprophylaxis? Estimation of adherence by an electronic pillbox. J Travel Med. 2006 Jan-Feb;13(1):8-14. doi: 10.1111/j.1708-8305.2006.00005.x. PMID 16412104
- [Background] Senn N, D'Acremont V, Landry P, Genton B. Malaria chemoprophylaxis: what do the travelers choose, and how does pretravel consultation influence their final decision. Am J Trop Med Hyg. 2007 Dec;77(6):1010-4. PMID 18165513
- [Background] Hatz C, Soto J, Nothdurft HD, Zoller T, Weitzel T, Loutan L, Bricaire F, Gay F, Burchard GD, Andriano K, Lefevre G, De Palacios PI, Genton B. Treatment of acute uncomplicated falciparum malaria with artemether-lumefantrine in nonimmune populations: a safety, efficacy, and pharmacokinetic study. Am J Trop Med Hyg. 2008 Feb;78(2):241-7. PMID 18256423
- [Background] Visser BJ, Wieten RW, Kroon D, Nagel IM, Belard S, van Vugt M, Grobusch MP. Efficacy and safety of artemisinin combination therapy (ACT) for non-falciparum malaria: a systematic review. Malar J. 2014 Nov 26;13:463. doi: 10.1186/1475-2875-13-463. PMID 25428624
- [Background] Voumard R, Berthod D, Rambaud-Althaus C, D'Acremont V, Genton B. Recommendations for malaria prevention in moderate to low risk areas: travellers' choice and risk perception. Malar J. 2015 Apr 1;14:139. doi: 10.1186/s12936-015-0654-y. PMID 25889529
- [Background] Schlagenhauf P, Petersen E. Standby emergency treatment of malaria in travelers: experience to date and new developments. Expert Rev Anti Infect Ther. 2012 May;10(5):537-46. doi: 10.1586/eri.12.42. PMID 22702318
- [Background] Jelinek T, Amsler L, Grobusch MP, Nothdurft HD. Self-use of rapid tests for malaria diagnosis by tourists. Lancet. 1999 Nov 6;354(9190):1609. doi: 10.1016/s0140-6736(99)01969-8. PMID 10560678
- [Background] Maltha J, Gillet P, Heutmekers M, Bottieau E, Van Gompel A, Jacobs J. Self-diagnosis of malaria by travelers and expatriates: assessment of malaria rapid diagnostic tests available on the internet. PLoS One. 2013;8(1):e53102. doi: 10.1371/journal.pone.0053102. Epub 2013 Jan 2. PMID 23301027
- [Background] Maltha J, Gillet P, Jacobs J. Malaria rapid diagnostic tests in travel medicine. Clin Microbiol Infect. 2013 May;19(5):408-15. doi: 10.1111/1469-0691.12152. Epub 2013 Feb 1. PMID 23373854